CLINICAL TRIAL: NCT07166510
Title: Reducing Burnout in Caregivers Through Yoga and Square Breathing Practices
Brief Title: Reducing Burnout in Healthcare Workers Through Yoga and Square Breathing Practices
Acronym: RESPYR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2025-A00849-40
Record Dates: First submitted 2025-09-03; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Burn-Out
Keywords: yoga; square breathing; emergency department
MeSH Terms: conditions — Burnout, Psychological; Emergencies | interventions — Yoga; Meditation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Emergency departement staff (Other): Emergency departement staff (nursing assistant, paramedic, medical dispatch assistant, registered nurse, physician)
  Interventions: Other: Yoga and meditation

INTERVENTIONS:
Other: Yoga and meditation — For 12 months, with no restrictions or imposed frequency, as often as the participant feels the need. They can take individual or group video-guided 15-minute breaks to do tailored yoga exercises targeting areas affected by repetitive movements, fatigue, and stress (hands, wrists, shoulders, and back), or mindfulness meditation sessions focused on managing fatigue, transitioning at the end of a shift, and post-shock relaxation.

SUMMARY:
The mental health of healthcare workers, burnout, and the resulting suicides are now described as a real "public health crisis." Emergency departments are not spared by this phenomenon; in fact, up to 71% of emergency physicians suffer from burnout. All professions are affected, with 49.2% of nurses reportedly affected by this phenomenon, and this figure rises to 90.7% of nursing assistants and 30% of paramedics providing advanced life support. However, ensuring the safety and protecting the physical and mental health of workers is a legal obligation in France.

In their latest recommendation on human factors in critical situations, SFAR experts suggest "limiting the factors responsible for burnout among caregivers exposed to crisis situations in order to reduce the risk of errors and unprofessional behavior." To achieve this, the importance of taking breaks in emergency medicine is already well recognized, and it is recommended that participants be given permission to take care of themselves through an agreement negotiated with peers and other staff members.

Furthermore, for several years now, the benefits of yoga in managing stress among healthcare workers seem to have been confirmed. Yoga is effective in reducing depression and anxiety, and it also improves sleep and clinical performance. It has also been shown to significantly reduce scores on the depersonalization and personal accomplishment items of the Maslach Burnout Inventory (MBI).

In addition, mindfulness meditation (MPC), based in particular on various breathing techniques including square breathing, is increasingly being studied, and SFAR experts suggest, with the help of these methods in particular, that "healthcare teams faced with critical situations benefit from psychological preparation for stress management to improve their experience and performance in such critical situations." Sudarshan Kriya Yoga, a technique that focuses primarily on breathing rhythm, has also been shown to be effective in improving well-being and reducing burnout among physicians.

Finally, yoga and mindfulness meditation administered together are effective in reducing stress and anxiety among healthcare workers, giving them greater attention, alertness, and ability to manage the stressful demands of work.

However, the combination of these two techniques through the implementation of video-guided breaks combining both techniques has never been studied.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18 or over
* Subjects who have been working for at least one year in the emergency department/emergency medical service/mobile emergency and resuscitation service of the selected centers as a nursing assistant, paramedic, medical dispatch assistant, registered nurse, or doctor
* Subjects who are affiliated with or beneficiaries of a social security system
* Consent signed by the participant regarding their participation in the study

Exclusion Criteria:

* Physical or psychological contraindications to practicing yoga or mindfulness meditation.
* Subjects who reported having been on sick leave for at least three months due to burnout prior to inclusion in the study
* Subjects who reported currently being monitored and/or treated by a healthcare professional for burnout
* Subjects who reported practicing yoga or meditation regularly (more than one day per week over the last three months)
* Scheduled absence of at least 3 months (e.g., maternity leave, availability, etc.)
* Subjects who did not wish to participate in the study.
* People benefiting from enhanced protection, namely minors, people deprived of their liberty by a judicial or administrative decision, people staying in a health or social care facility, and adults under legal protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the impact after 6 months of implementing breaks consisting of 15-minute video-guided yoga or meditation sessions on burnout among emergency department staff at participating centers. | 6 months
  Proportion of participants experiencing burnout at 6 months, compared to inclusion.
  Burnout is defined as a high score on the emotional exhaustion scale (≥27) and either: a high score on the depersonalization scale (≥10), or a low score on the personal accomplishment scale (≤33), according to the standard thresholds of the Maslach Burnout Inventory (MBI-HSS).

SECONDARY OUTCOMES:
Assess the change in the proportion of participants experiencing burnout at 3 months (M3) and 12 months (M12), using the same composite definition as that used for the primary endpoint. | 3 months and 12 months
  Proportion of participants experiencing burnout at 3 months and 12 months, according to the same composite definition as for the primary endpoint
Explore the evolution of continuous scores for the three dimensions of burnout (emotional exhaustion, depersonalization, personal accomplishment), measured by the MBI-HSS, between inclusion (T0), 3 months, 6 months, and 12 months. | From enrollment to 12 months
  Changes in continuous scores obtained on each of the three subscales of the Maslach Burnout Inventory (emotional exhaustion, depersonalization, personal accomplishment) between inclusion (T0), 3 months, 6 months, and 12 months.
Assess the impact of the intervention on participants' quality of life, via changes in SF-12 mental and physical scores collected at baseline, then at 3, 6, and 12 months. | From enrollment to 12 months
  Changes in average scores obtained on the physical and mental components of the SF-12 between inclusion, 3 months, 6 months, and 12 months.
Assess adherence to the program, based on the initial participation rate and the persistence rate until the end of the study, among healthcare personnel in the emergency departments of participating centers. | From enrollment to 12 months
  Initial participation rate, defined as the number of participants who agreed to participate in the study relative to the total number of eligible professionals.
  Effective participation rate, defined as the number of participants who continued the intervention until the end of the study relative to the number of participants initially included.

CONTACTS AND LOCATIONS:
Overall Officials: Céline ABONNEAU, Project Manager, Study Chair — Poitiers University Hospital
Locations (2):
- France (2):
  - Bordeaux University Hospital, Bordeaux
  - Poitiers University Hospital, Poitiers

IPD SHARING:
Plan to Share IPD: No